CLINICAL TRIAL: NCT07199348
Title: A Safety and Performance Study of the Use of EmboBio for the Intra-arterial Treatment of Abdominopelvic Bleeding: EMBOBIO-1
Brief Title: A Safety and Performance Study of the Use of EmboBio for the Intra-arterial Treatment of Abdominopelvic Bleeding
Acronym: EMBOBIO-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Embobio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00222-47; 2025-A00222-47 (Other: ANSM)
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Abdomino-pelvic Surgery; Bleeding; Embolization
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embobio (Experimental): Patient implanted with Embobio
  Interventions: Device: Embobio

INTERVENTIONS:
Device: Embobio — Embolization with the device Embobio

SUMMARY:
This research conducted by EMBOBIO SAS is intended for patients with bleeding or at risk of bleeding in the abdominal-pelvic region requiring embolization.

The EmboBio device (embolization implant) is a Class IIb medical device that is not CE marked (meaning that it is not yet commercially available on the European market).

The objective of the study is to demonstrate the safety and performance of the EmboBio medical embolization device in humans in order to obtain CE marking, the European authorization required for the commercialization of medical devices.

Safety will be assessed by collecting data on events that may be related to the device, and the device will be considered effective if the target arteries are completely occluded (blocked) at the end of the operation.

The plan is to include 45 patients (men and women aged 18 or over who have given their consent to participate in the study) requiring embolization in the abdominal-pelvic region in French hospitals over a period of 12 months. The patient's full participation is requested for a period of approximately 6 months.

DETAILED DESCRIPTION:
Abdominopelvic bleeding may occur in different and various circumstances, in a spontaneous way, after a trauma, in a neoplasic context, after a visceral aneurysm's rupture, during or after a surgical treatment. They require fast and effective treatment, as they can be rapidly life-threatening, and that's where embolization steps in.

Embolization is a recent interventional radiology technique whose objective is the occlusion of arterial or venous vessels. Unlike so-called conventional surgical techniques, it is a minimally invasive treatment consisting in endovascular navigation using catheters and microcatheters to reach target vessels where the embolic agent is delivered. The choice of the embolic agent is guided by the indication of the procedure as well as the embolization site. Available permanent embolic agents include calibrated microparticles, metallic implants (coils, plugs) and bioglue. Although the ideal embolic agent does not exist, the choice of material remains a fundamental step in embolization procedures, and the development of new agents is an important avenue of research.

The choice of the embolic agent for bleeding control is based on the site of bleeding, the size of the artery, how fast the bleeding can be controlled but also the time required for embolic agent preparation, its price and the physician's preference. In this indication, the most often used permanent embolic agents are coils. Known adverse device effects of coils are risks of migration, non-target embolization, infection and damage to the wall vessels.

With the urgency of climate change and the demand for natural products in reaction to the overconsumption of chemicals for decades, both food and health industries have experienced a very strong demand for products with a biological process, both respectful of the environment in its design, and of the organism in its distribution. In this context, it seems appealing and important to develop new agents designed from new materials. Indeed, the use of organic materials is a game-changer that is both innovative and promising. More than these aspects, the development of organic embolic material seems necessary to improve the biocompatibility of implantable medical devices with the organism.

To conclude, the best embolic agent for abdominopelvic bleeding should provide a fast and effective long-term occlusion of the bleeding arteries, be safe, prepared speedily, easy to use, cheap and ecofriendly.

Embobio has been designed and developed to meet all these expectations. Embobio is the first organic agent designed for permanent embolization. We demonstrated in a preclinical study that this new agar-agar embolization implant is easy to use and effective in stopping bleeding in a hemorrhagic shock model, making it well-suited for emergency interventional radiology procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient presenting with an arterial abdominopelvic bleeding or risk of bleeding requiring embolization with a permanent embolic agent, i.e. abdominal solid organs hemorrhage including angiomyolipoma, visceral aneurysms and pseudoaneurysms actively bleeding or at risk of bleeding (upper or lower gastrointestinal arteries), pelvic hemorrhage, postpartum hemorrhage in case of active leakage visualized by contrast media extravasation, soft tissue hemorrhage
* Patient having provided a written informed consent

Exclusion Criteria:

* Known hypersensitivity to Agar-Agar
* Known hypersensitivity to iodinated contrast media
* Patient unable or unwilling to provide a written informed consent
* Patient unable to provide informed consent due to his clinical condition
* Patient participating in another interventional study
* Patient implanted with Embobio device at a previous operating time
* Vulnerable, pregnant, and breastfeeding population
* Patient unwilling or unable to follow the study schedule
* Patients unable to receive prior information on the clinical investigation due to the urgency of the situation
* Target arteries diameter > 2 mm
* Vascular anatomy preventing proper placement of the catheter.
* Arteriovenous shunts with a high flow rate or a diameter greater than 2 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Adverse Device Effects (SADE) | 24 hours
  The primary endpoint of the pilot stage is the rate of SADE (serious adverse events, probably or certainly related to investigational device deficiencies) within 24 hours.
Rate of technical success | At the end of the procedure
  The primary performance endpoint is the technical success defined by the successful achievement of embolization of the target artery/arteries, and the absence of extravasation of contrast of target artery/arteries after arterial embolization at the end of the procedure.
Description of procedural data : dosimetry | At the end of the procedure
  Dosimetry data during the procedure
Description of procedural data : quantity of Embobio | At the end of the procedure
  Quantity of Embobio used for embolization
Description of procedural data : time to bleeding control | At the end of the procedure
  Time needed to control the bleeding
Description of procedural data : procedure duration | At the end of the procedure
  Total duration of the procedure

SECONDARY OUTCOMES:
Rate of adverse events and adverse device effects | 1 week
  The rate of adverse events, serious adverse events and adverse device effects, up to 1 week.
Rate of immediate clinical success | At the end of the procedure
  Immediate clinical success will be defined as the successful achievement of embolization, and the absence of extravasation of contrast after arterial embolization at the end of the procedure
Rate of clinical success | 7 days
  Clinical success will be defined as the absence of rebleeding of target artery(ies) requiring reintervention (repeat embolization or additional surgery) within 7 days.
Mortality rate | 7 days
  Mortality rate related to device use, embolization procedure and pathology at 7 days
Name and number of the potentiel other devices used to achieve occlusion | At the end of the procedure
  Name and number of the devices used to achieve occlusion (other than Embobio) and whether their use was anticipated or due to investigational device failure.
Interventional Radiologist's satisfaction questionnaire | At the end of the procedure
  (translated from French) Q1. Did you achieve the expected embolization results?
  * Yes
  * Partially
  * No
  Q2. How would you rate the ease of handling Embobio?
  * Difficult
  * Average
  * Easy
  * Very easy
  Q3. How would you describe the ease of injection?
  * Very good
  * Good
  * Average
  * Poor
  Q4. How do you find the speed of occlusion?
  * Very good
  * Good
  * Average
  * Poor
  Q5. How do you find the use of Embobio compared to other agents (coils, particles)?
  * More difficult
  * Equivalent
  * Easier

IPD SHARING:
Plan to Share IPD: No